CLINICAL TRIAL: NCT05588284
Title: Effect of Endovascular Thrombectomy for Femoral Popliteal Vein Thrombosis on Venous Valve Function Maintenance: a Single-center, Single-arm Prospective Observational Study
Brief Title: Preservation of Venous Valvular Function After PMT for Acute DVT
Acronym: PREFER
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Kaichuang Ye, MD, PhD, Vice professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAL03
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute Deep Venous Thrombosis of Femoral Vein (Disorder)
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pharmacomechanical Catheter-directed Thrombolysis for acute DVT (Experimental): AngioJet, Boston Scientific
  Interventions: Device: AngioJet device
- anticoagulation alone for acute DVT (Placebo Comparator): anticoagulation alone for acute DVT
  Interventions: Other: anticoagulation alone

INTERVENTIONS:
Device: AngioJet device — A device can be used for thrombus aspiration and thrombolysis.
  Other Names: Zalente
  Arms: Pharmacomechanical Catheter-directed Thrombolysis for acute DVT
Other: anticoagulation alone — a medicine for anticoagulation therapy
  Other Names: rivaroxaban
  Arms: anticoagulation alone for acute DVT

SUMMARY:
To evaluate the venous valvular function after pharmacomechanical thrombectomy (PMT) for acute femoral-popliteal venous thrombosis.

DETAILED DESCRIPTION:
All patients presenting with symptoms in the lower extremity due to the femoral venous thrombosis involving or not involving iliac and popliteal veins treated with percutaneously pharmacomechanical catheter-directed thrombolysis via AngioJet devices or anticoagulation alone were included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute symptomatic proximal DVT involving the femoral, and/or popliteal vein, common femoral vein, iliac veins (with or without other involved ipsilateral veins) were enrolled at seven vascular centers in China. Patients were treated with PCDT via Zelante device (Boston Scientific).

Exclusion Criteria:

* Participants were excluded if they had symptoms for more than 14 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Valvular reflux prevalence | at 12 months after procedure
  Proportion of patients with femoral venous valve reflux at 1 year after procedure

SECONDARY OUTCOMES:
Cumulative Incidence of Post-Thrombotic Syndrome (Villalta Scale) | at 6, 12 and 24 months after procedure
  Patients who experienced one of the following occurrences in the index leg between the 12 month and 24 month post-randomization follow-up visits, inclusive: 1) Villalta score of 5 or greater; 2) leg ulcer; or 3) late endovascular procedure performed to treat severe venous disease. The Villalta scale ranges from 0-33 points, with higher scores being worse.
Patency rate of femopopliteal vein and iliofemoral vein | at 6, 12 and 24 months after procedure
  Patients who presented with patent femopopliteal vein and iliofemoral vein

CONTACTS AND LOCATIONS:
Overall Officials: Kaichuang Ye, MD, PhD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (7):
- China (7):
  - Chuzhou People's Hospital, Chuzhou, Anhui
  - Center hospital of Putu, Shanghai, Shanghai Municipality
  - Central Hospital of Songjiang, Shanghai, Shanghai Municipality
  - North Branch of Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Fengchen Hospital, Shanghai, Shanghai Municipality
  - Taizhou Municipal hospital, Taizhou, Zhejiang